CLINICAL TRIAL: NCT04688008
Title: An Open-label, Randomized, Single-dose, Two -Period, Crossover Study to Investigate the Relative Bioavailability of Early Phase and Late Phase Hetrombopag Olamine Formulations in Healthy Chinese Adult Subjects Under Fasting Conditions.
Brief Title: Relative Bioavailability of Early Phase and Late Phase Hetrombopag Olamine Formulations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SHR8735-112
Record Dates: First submitted 2020-12-11; First posted 2020-12-29 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2020-12

CONDITIONS: Bioavailability Study
MeSH Terms: interventions — hetrombopag

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment sequence #1 (Other): 29 of 58 subjects were given single oral dose of early phase hetrombopag olamine formulation in period 1 and late phase formulation in period 2
  Interventions: Drug: Hetrombopag
- Treatment sequence #2 (Other): 29 of 58 subjects were given single oral dose of late phase hetrombopag olamine formulation in period 1 and early phase formulation in period 2
  Interventions: Drug: Hetrombopag

INTERVENTIONS:
Drug: Hetrombopag — Drug: Early phase hetrombopag olamine formulation single oral dose of 5 mg hetrombopag under fasting conditions
  Drug: Late phase hetrombopag olamine formulation single oral dose of 5 mg hetrombopag under fasting conditions

SUMMARY:
The primary objective of the study is to evaluate the relative bioavailability of early phase and late phase hetrombopag olamine formulations in healthy Chinese adult subjects under fasting conditions. The secondary objective of the study is to evaluate the safety of hetrombopag olamine in healthy Chinese adult subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent before the trial, and fully understand the trial content, process and possible adverse reactions;
2. Ability to complete the study as required by the protocol;
3. Healthy male or female subjects aged 18 to 45 (including 18 and 45) at the date of signing the informed consent;
4. Body mass index (BMI) within the range of 19 ~ 26 kg /m2 (including 19 and 26);

Exclusion Criteria:

1. Allergic constitution;
2. History of drug use, or drug abuse screening positive;
3. Alcoholic or often drinkers;
4. History of deep vein thrombosis, or any other thromboembolic event;
5. A clear medical history of important primary organ diseases such as nervous system, cardiovascular system, urinary system, digestive system, respiratory system, metabolism and musculoskeletal system.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2020-09-18 (Actual); Primary Completion 2020-10-12 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Peak plasma concentration (Cmax) | 0-120 hours post dose
Area Under the plasma concentration vs time curve (AUC0-120). | 0-120 hours post dose
area under the blood concentration vs time curve (AUC0-inf). | 0-infinity

SECONDARY OUTCOMES:
Time to Reach Maximum Drug Concentration in Plasma After Single Dose (Tmax) | 0-120 hours post dose
Half-life Associated With the Terminal Slope (t½) | 0-120 hours post dose

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Hospital of Anhui Medical University, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No